CLINICAL TRIAL: NCT04495777
Title: Prevalence of Temporomandibular Disorders and Its Association With Oral Parafunctions, Neck Pain and Function in Female Turkish Healthcare Students: A Cross-Sectional Study
Brief Title: Prevalence of Temporomandibular Disorders and Its Association With Oral Parafunctions, Neck Pain and Function
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, GulOznur KARABICAK, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: tmd_101
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Temporomandibular Disorder; Neck Pain
Keywords: temporomandibular; students; prevalence; parafunctional habit; neck pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: students were assessed in order to have a risk for TMD in order to their status of having parafunctional habits and neck pain
  Interventions: Other: Fonseca Anamnestic Index

INTERVENTIONS:
Other: Fonseca Anamnestic Index — Fonseca Anamnestic Index was developed to assess the severity of temporomandibular disorders, based on its signs and symptoms. It has been proposed as a low cost and easy to apply alternative and has been used in screening for TMD in a non-patient population5. It was created with 10 items with 3 options of answers (specific scores): "yes (10 points)", "sometimes (5 points)" and "no (0 points)". The final score of the instrument is determined by the sum of the scores of all items, allowing the following classifications: the absence of signs and symptoms of TMD (0-15 points), mild TMD (20-45 points), moderate TMD (50-65 points), and severe TMD (70-100 points) (19).

SUMMARY:
Purpose: To determine the prevalence of temporomandibular disorders (TMD) in female healthcare students and to assess its association with oral parafunctions, neck pain and function.

Methods: Female medical students will be included in the study on a voluntary basis using stratified sampling method according to the department they were being educated. The presence and severity of TMD will be assessed with the Fonseca's Anamnestic Index (FAI). The oral parafunctions will be self-reported with the Oral Behavior Checklist (OBC). The neck pain and function will be recorded with the Core Outcome Measure Index (COMI). A Chi-square test and Spearman correlation analysis will used for statistical analysis.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) has a multifactorial etiology related to parafunctional habits, emotional and psychological factors, trauma, posture, other musculoskeletal, or rheumatic disorders (1). Symptoms of TMD may include temporomandibular joint pain and clicks, headache, myofascial pain, decreased mandibular range of motion, masticatory muscle fatigue, limitation of mouth opening, pain when chewing, tinnitus, neuralgias, and bruxism (1,2). The severity of symptoms is related to the age and gender of the patients. Women showed a higher prevalence of TMD symptoms, with proportions varying from two to six women for each man, usually with ages between 20 and 40 years3. The distribution of age and gender in TMD, suggests a possible link between its pathogenesis and the female sex hormone, the estrogen, or between TMD and the mechanisms of pain modulation, as women show more sensitivity to most of the pain modalities (3,4) Epidemiologic studies showed that TMD prevalence in the students ranges from 50% to 77% (5-7). Several studies reported that a higher prevalence of TMD ranges from 47% to 81% in the Turkish student population (8-13). However, in some cases especially in students, the presence of TMD is asymptomatic. Therefore, the diagnosis of early symptoms and signs of TMD is crucial in preventing or minimizing TMD signs and symptoms (9).

Parafunctional habits such as bruxism, tooth clenching, gum chewing, biting foreign objects, and prolonged nail-biting might increase the risk of developing TMD (14). Even there are several studies examining the association of TMD and oral parafunctions in students (15-17); still, more studies are need to identify which oral behaviors cause TMD patients and healthy populations (18). Therefore, understanding the TMD symptoms in association with the oral parafunctions could provide different perspectives and an efficient treatment program (15).

To our knowledge, there is no study about TMD prevalence in female healthcare students and its association with oral parafunctions, neck pain, and function. The aims of this cross-sectional study were: (1) to evaluate the prevalence of TMD in female healthcare students and (2) to determine the association of TMD severity with oral parafunctional habits, neck pain and function.

ELIGIBILITY:
Inclusion Criteria:

* be Adnan Menderes University student
* female gender
* express consent to participate voluntarily in the study

Exclusion Criteria:

* with recent trauma to head and face,
* history of systematic diseases and neurological disorders
* currently an ongoing orthodontic treatment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — students who define themselves as female are included in our study
Study Population: University students who are currently ongoing their education in healthcare department
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index | baseline
  Fonseca Anamnestic Index was developed to assess the severity of temporomandibular disorders, based on its signs and symptoms. It has been proposed as a low cost and easy to apply alternative and has been used in screening for TMD in a non-patient population5. It was created with 10 items with 3 options of answers (specific scores): "yes (10 points)", "sometimes (5 points)" and "no (0 points)". The final score of the instrument is determined by the sum of the scores of all items, allowing the following classifications: the absence of signs and symptoms of TMD (0-15 points), mild TMD (20-45 points), moderate TMD (50-65 points), and severe TMD (70-100 points) (19).

SECONDARY OUTCOMES:
Oral parafunction | baseline
  Oral behaviors checklist is a self-report questionnaire for determining the frequency of oral parafunctional behaviors which are any abnormal behavior or functioning of the oral structures and associated muscles in the past one month. Original questionnaire consists of 21items, 2 items for oral behaviors during sleep, and 19 items for oral behaviors during waking hours. In this study the questionnaire was modified and two of the questions were exctracted due to study of Hayek et al25. Each item is scored from 0-4 based on the frequency of activity performed: a score of 0=none of the time; a score of 1=a little of the time; a score of 2=some of the time; a score of 3=most of the time and score of 4=all the time; with a range of 0-76 18.The sum of scoring had the following scheme: none = 0, low = 1-16, and high = 17-76 (20).
Neck pain and function | baseline
  The COMI-neck is a short, self-administered outcome instrument consisting of just seven items to evaluate the five dimensions pain, neck-related function, symptom-specific well-being, general quality of life, and disability (social and work) (21,22). The two pain items use a 0-10 graphic rating scale; all other items use a 5-point adjective scale. For COMI summary score, each of the domain scores is transformed to a 0-10 scale and these are then averaged to give a score ranging from 0 to 10, with higher scores indicating a worse status (23).

CONTACTS AND LOCATIONS:
Overall Officials: Gul Oznur KARABICAK, Phd, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Gul Oznur KARABICAK, Aydin, Turkey (Türkiye)

REFERENCES:
- [Background] Pedroni CR, De Oliveira AS, Guaratini MI. Prevalence study of signs and symptoms of temporomandibular disorders in university students. J Oral Rehabil. 2003 Mar;30(3):283-9. doi: 10.1046/j.1365-2842.2003.01010.x. PMID 12588501
- [Background] Kuc J, Szarejko KD, Sierpinska T. Evaluation of Orofacial and General Pain Location in Patients With Temporomandibular Joint Disorder-Myofascial Pain With Referral. Front Neurol. 2019 May 29;10:546. doi: 10.3389/fneur.2019.00546. eCollection 2019. PMID 31191438
- [Background] Schmid-Schwap M, Bristela M, Kundi M, Piehslinger E. Sex-specific differences in patients with temporomandibular disorders. J Orofac Pain. 2013 Winter;27(1):42-50. doi: 10.11607/jop.970. PMID 23424719
- [Background] Nekora-Azak A, Evlioglu G, Ceyhan A, Keskin H, Berkman S, Issever H. Estrogen replacement therapy among postmenopausal women and its effects on signs and symptoms of temporomandibular disorders. Cranio. 2008 Jul;26(3):211-5. doi: 10.1179/crn.2008.028. PMID 18686498
- [Background] Nomura K, Vitti M, Oliveira AS, Chaves TC, Semprini M, Siessere S, Hallak JE, Regalo SC. Use of the Fonseca's questionnaire to assess the prevalence and severity of temporomandibular disorders in Brazilian dental undergraduates. Braz Dent J. 2007;18(2):163-7. doi: 10.1590/s0103-64402007000200015. PMID 17982559
- [Background] Karthik R, Hafila MIF, Saravanan C, Vivek N, Priyadarsini P, Ashwath B. Assessing Prevalence of Temporomandibular Disorders among University Students: A Questionnaire Study. J Int Soc Prev Community Dent. 2017 Jun;7(Suppl 1):S24-S29. doi: 10.4103/jispcd.JISPCD_146_17. Epub 2017 Jun 20. PMID 28713764
- [Background] Lung J, Bell L, Heslop M, Cuming S, Ariyawardana A. Prevalence of temporomandibular disorders among a cohort of university undergraduates in Australia. J Investig Clin Dent. 2018 Aug;9(3):e12341. doi: 10.1111/jicd.12341. Epub 2018 Mar 31. PMID 29604182
- [Background] Emel Dervis N. Prevalence of Temporomandibular Disorder in Turkish University Students: a Questionnaire Study. Balk J Dent Med. 2019; 23 (2): 80-87 doi:10.2478/bjdm-2019-0015
- [Background] Türken R, Büyük SK, Yaşa Y. Diş Hekimliği Fakültesi Öğrencilerinde Temporomandibular Eklem Rahatsızlıklarının ve Ağız Sağlığı Alışkanlıklarının Değerlendirilmesi. Acıbadem Üniversitesi Sağlık Bilim Derg. 2020;11(2):208-213. https://doi.org/10.31067/0.2018.83.
- [Background] Tanhan A, Yıldız A, Demirbüken İ, Polat MG. Sağlık Bilimleri Öğrencilerinde Temporomandibular Eklem Disfonksiyon Riskinin Araştırılması. Sak Med J. 2019. doi:10.31832/smj.490740
- [Background] Yalcin Yeler D, Yilmaz N, Koraltan M, Aydin E. A survey on the potential relationships between TMD, possible sleep bruxism, unilateral chewing, and occlusal factors in Turkish university students. Cranio. 2017 Sep;35(5):308-314. doi: 10.1080/08869634.2016.1239851. Epub 2016 Oct 6. PMID 27707365
- [Background] Ozdinc S PhD, Ata H MSc, Selcuk H MSc, Can HB MSc, Sermenli N MSc, Turan FN PhD. Temporomandibular joint disorder determined by Fonseca anamnestic index and associated factors in 18- to 27-year-old university students. Cranio. 2020 Sep;38(5):327-332. doi: 10.1080/08869634.2018.1513442. Epub 2018 Sep 8. PMID 30198391
- [Background] Ayalı A, Ramoğlu S. KUZEY KIBRIS'TA DİŞ HEKİMLİĞİ FAKÜLTESİ ÖĞRENCİLERİNDE TEMPOROMANDİBULER EKLEM DİSFONKSİYONU'NUN PREVALANSI. Atatürk Üniversitesi Diş Hekim Fakültesi Derg. 2015;24(3). doi:10.17567/dfd.91850
- [Background] Oliveira LK, Almeida Gde A, Lelis ER, Tavares M, Fernandes Neto AJ. Temporomandibular disorder and anxiety, quality of sleep, and quality of life in nursing professionals. Braz Oral Res. 2015;29:S1806-83242015000100265. doi: 10.1590/1807-3107BOR-2015.vol29.0070. PMID 26039910
- [Background] Chatzopoulos GS, Sanchez M, Cisneros A, Wolff LF. Prevalence of temporomandibular symptoms and parafunctional habits in a university dental clinic and association with gender, age, and missing teeth. Cranio. 2019 May;37(3):159-167. doi: 10.1080/08869634.2017.1399649. Epub 2017 Nov 16. PMID 29143569
- [Background] Lovgren A, Osterlund C, Ilgunas A, Lampa E, Hellstrom F. A high prevalence of TMD is related to somatic awareness and pain intensity among healthy dental students. Acta Odontol Scand. 2018 Aug;76(6):387-393. doi: 10.1080/00016357.2018.1440322. Epub 2018 Feb 18. PMID 29457522
- [Background] Paduano S MD, DDS, Bucci R DDS, PhD, Rongo R DDS, PhD, Silva R DDS, Michelotti A DDS. Prevalence of temporomandibular disorders and oral parafunctions in adolescents from public schools in Southern Italy. Cranio. 2020 Nov;38(6):370-375. doi: 10.1080/08869634.2018.1556893. Epub 2018 Dec 14. PMID 30547719
- [Background] Leketas M, Saferis V, Kubilius R, Cervino G, Bramanti E, Cicciu M. Oral Behaviors and Parafunctions: Comparison of Temporomandibular Dysfunction Patients and Controls. J Craniofac Surg. 2017 Nov;28(8):1933-1938. doi: 10.1097/SCS.0000000000003945. PMID 28930927
- [Background] Bevilaqua-Grossi D, Chaves TC, de Oliveira AS, Monteiro-Pedro V. Anamnestic index severity and signs and symptoms of TMD. Cranio. 2006 Apr;24(2):112-8. doi: 10.1179/crn.2006.018. PMID 16711273
- [Background] Al Hayek SO, Al-Thunayan MF, AlGhaihab AM, AlReshaid RM, Omair A. Assessing stress associated with temporomandibular joint disorder through Fonseca's anamnestic index among the Saudi physicians. Clin Exp Dent Res. 2018 Dec 26;5(1):52-58. doi: 10.1002/cre2.157. eCollection 2019 Feb. PMID 30847233
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):367-73. doi: 10.1007/s00586-009-0942-8. Epub 2009 Mar 25. PMID 19319578
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective: part 2. Minimal clinically important difference for improvement and deterioration as measured with the Core Outcome Measures Index. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):374-9. doi: 10.1007/s00586-009-0931-y. Epub 2009 Mar 19. PMID 19296136
- [Background] Karabicak GO, Hazar Kanik Z, Gunaydin G, Pala OO, Citaker S. Reliability and validity of the Turkish version of the Core Outcome Measures Index for the neck pain. Eur Spine J. 2020 Jan;29(1):186-193. doi: 10.1007/s00586-019-06169-w. Epub 2019 Oct 31. PMID 31673855